CLINICAL TRIAL: NCT05593653
Title: Treating Insomnia and Improving Glycemic Control in Midlife Women With Insomnia and Pre-diabetes
Brief Title: Efficacy of Suvorexant in the Treatment of Insomnia in Midlife Women With Pre-Diabetes
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shadab A Rahman, Study Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022P000768
Record Dates: First submitted 2022-10-21; First posted 2022-10-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Insomnia; Diabetes; Menopause
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Diabetes Mellitus | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- suvorexant (Experimental): 20mg taken at bedtime for 4 weeks
  Interventions: Drug: Suvorexant
- placebo (Placebo Comparator): placebo taken at bedtime for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Suvorexant — 20mg taken at bedtime for 4 weeks
  Other Names: Belsomra
  Arms: suvorexant
Drug: Placebo — placebo taken at bedtime for 4 weeks
  Arms: placebo

SUMMARY:
The aim of this study is to determine if suvorexant can help treat the severity of insomnia in midlife women who are pre-diabetic.

DETAILED DESCRIPTION:
The purpose of this research study is to investigate if suvorexant can help treat the severity of insomnia (a chronic sleep disorder) in midlife women who are pre-diabetic, and to learn whether improvement in insomnia symptoms is linked with improvement in blood sugar levels. This is a double-blind, randomized placebo-controlled crossover trial. Study procedures are conducted over a 14-week period (2-week screening period, 4-week treatment period [Block 1], 4-week washout, and 4-week treatment period [Block 2]). During each treatment block, participants take a daily pill - during one block, they take suvorexant and during the other block, they take a placebo (randomized to the order). Primary data collection includes blood draws, monitoring glucose and lipid levels, actigraphy, questionnaires, and daily diaries.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women aged 40-65 years
* Postmenopausal or late perimenopausal
* Meets criteria for Insomnia Disorder
* Score on the Insomnia Severity Index (ISI) measure ≥15
* Subjective and sustained sleep disruption during screening
* Hot flashes present, including at night
* Pre-diabetic per guidelines from the American Diabetes Association

Exclusion Criteria:

* Diagnosis of other primary sleep disorders
* Shift worker
* Frequent use of hypnotic medications
* Unwillingness to refrain from taking any sleep medications during the study period
* Current major depressive episode
* Suicidal ideation
* Lifetime history of bipolar disorder, psychosis, or other serious mental health problem
* Current alcohol/substance use disorder
* Current or prior diagnosis of diabetes mellitus
* Use of an insulin sensitizer or a pharmacologic treatment for pre-diabetes
* Extreme obesity
* Current use of systemic hormonal therapies
* Renal or hepatic disease
* Pregnancy or breastfeeding
* Recent malignancy
* Recent surgery
* Neurological disorder or cardiovascular disease raising safety concerns
* Medical instability considered to interfere with study procedures
* Concomitant medications with drug interaction or co-administration concerns
* Contraindications or allergic responses to suvorexant
* Recent travel across time zones
* Excessive coffee or cigarette use
* Unwilling to limit alcohol, nicotine, and caffeine consumption during study

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 61 (Estimated)
Dates: Start 2023-01-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index Score | baseline to 4 weeks
  The Insomnia Severity Index (ISI) is a 7-item self-rated scale to assess the severity of insomnia symptoms. The total ISI score is the sum of all questions, with a total range from 0-28 with higher values indicating worse insomnia.

SECONDARY OUTCOMES:
Fasting Plasma Glucose | baseline to 4 weeks
  Fasting plasma glucose is determined from a blood sample collected at least 8 hours since last food intake. Range indications: 0-99 mg/dL is normal, 100-125 mg/dL is pre-diabetic, and 126 mg/dL+ indicates diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Shadab Rahman, PhD MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States